CLINICAL TRIAL: NCT03347851
Title: Investigation of Post-surgical Aortic Hemodynamics After Aortic Valve Replacement
Brief Title: Post-surgical Aortic Hemodynamics After Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: CryoLife, Inc. (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Organization: CryoLife (Unknown)
Other Study IDs: 2017-1
Record Dates: First submitted 2017-10-24; First posted 2017-11-20 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Valve Heart Disease
Keywords: mechanical heart valve; On-X
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- On-X AAP: Patients with prior AVR surgery with the CryoLife On-X Ascending Aortic Prosthesis (AAP).
  Interventions: Other: MRI; Other: Transthoracic echocardiography exam
- SJM Masters or Carbomedics Carbo-seal: Patients with St. Jude Medical Masters HP Valved Graft with Gelweave Valsalva™ Technology or Carbomedics Carbo-seal (including Carbo-seal Valsalva) mechanical aortic valve prostheses patients
  Interventions: Other: MRI; Other: Transthoracic echocardiography exam

INTERVENTIONS:
Other: MRI — Enrolled patients will complete a non-contrast cardiac MRI
Other: Transthoracic echocardiography exam — Enrolled patients will complete a transthoracic echocardiography exam.

SUMMARY:
The purpose of this pilot study is to obtain both near valve and downstream flow characteristics, using 3D transthoracic echocardiography and 4D flow MRI respectively, in an existing patient population at Northwestern Memorial Hospital, to determine the hinge washout characteristics and downstream flow patterns of the On-X valve and compared to competing designs.

DETAILED DESCRIPTION:
Prospective, concurrent 4D flow Magnetic Resonance Imaging (MRI) and echocardiography of On-X and St Jude Medical (SJM) Masters HP or Carbomedics Carbo-seal or Carbo-seal Valsalva aortic valve replacement (AVR) patients will be performed. Echocardiography analysis will include: valve function (opening angle), pressure gradients, and degree of valve washout. MRI analysis will focus on downstream flow patterns (helicity and vorticity), energy loss, pressure recovery, and measurement of wall shear stress in the anastomosis regions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18-89 years of age
* Patients with aortic valve disease who within the last five years underwent AVR using the On-X aortic valve, SJM Masters HP, or Carbomedics aortic valves.

Exclusion Criteria:

* Patients contraindicated against MRI
* Patients with pacemakers, cochlear (in the ear) implants, or aneurysm clips or patients who have worked with metal
* Patients unwilling or unable to give written informed consent
* Pregnant women
* Prisoners
* Patients with an Effective Orifice Area index (EOAi) <0.85 cm2/m2

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic valve disease who within the last five years underwent AVR using the On-X aortic valve, SJM Masters HP, or Carbomedics aortic valves.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Downstream flow patterns (helicity and vorticity) | 3 months
  MRI data analysis; Helicity and vorticity graded (1-3) by blinded reviewers.
Hinge washout | 3 months
  MRI data analysis; Yes/No
Energy loss | 3 months
  MRI data analysis; Irreversible energy loss quantified.Efforts will include the quantification of turbulent kinetic energy. This is representative of permanent pressure loss.
Wall shear stress (WSS) | 3 months
  MRI data analysis; WSS, the tangential force exerted by blood flow on the vessel wall, measured in the anastomosis regions

SECONDARY OUTCOMES:
Ejection Fraction (%) | 3 months
Primary EDV (ml) | 3 months
  End Diastolic Volume
Normalized EDV (ml/m^2) | 3 months
  End Diastolic Volume
Primary ESV (mL) | 3 months
  End Systolic Volume
Normalized ESV (mL/m^2) | 3 months
  End Systolic Volume
Peak Velocity (m/s) | 3 months
Mean velocity (m/s) | 3 months
Peak transvalvular pressure gradient (mmHg) | 3 months
Mean transvalvular pressure gradient (mmHg) | 3 months
Effective Orifice Area (EOA) | 3 months
Effective Orifice Area index (EOAi) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States